CLINICAL TRIAL: NCT00827346
Title: Platelet Function Monitoring in Patients Treated With Clopidogrel at the Time of Primary Percutaneous Coronary Angioplasty
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Michel Le May, UOHI
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: MRL-A2; 2008239-01H
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Platelet Reactivity
MeSH Terms: interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Active Comparator): 600-mg double dose
  Interventions: Drug: Clopidogrel
- Group 2 (Active Comparator): 600/600-mg double loading dose (first dose 600 mg given immediately upon arrival at the hospital and the second dose 600 mg, 3 hours after the first loading dose for a total of 900 mg
  Interventions: Drug: Clopidogrel
- Group 3 (Active Comparator): Clopidogrel 900mg
  Interventions: Drug: Clopidogrel
- Group 4 (Active Comparator): First dose 600 mg given immediately upon arrival at the hospital and the second dose 300 mg, 3 hours after the first loading dose for a total of 900 mg
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 600 mg now
  Arms: Group 1
Drug: Clopidogrel — 600 mg now and 600 mg in 3 hours
  Arms: Group 2
Drug: Clopidogrel — 900 mg now
  Arms: Group 3
Drug: Clopidogrel — 600 mg now and 300 mg in 3 hours
  Arms: Group 4

SUMMARY:
Platelets are a major component of clot formation which can lead to clotting events such as heart attack. During treatment for a heart attack, doctors try to remove this blockage as quickly as possible so that the heart can recover and start to work properly again. The standard of care at the Heart Institute for patients having a heart attack is a procedure called a Percutaneous Coronary Angioplasty. A drug called Clopidogrel (Plavix) is routinely used prior to the angioplasty to prevent blood clots. Patients usually remain on Clopidogrel for at least one year following the angioplasty. Clopidogrel works by preventing the blood from forming sticky substances called platelets, which clump together to form clots. Despite the routine use of Clopidogrel, some patients still return to the hospital with another heart attack, or with more chest pain. There is a growing body of evidence that recurrence of these complications may be attributed to some patients having a poor response to Clopidogrel.

This pilot study will examine how platelets react to different doses of Clopidogrel given to patients having a heart attack.

DETAILED DESCRIPTION:
Platelets are a major component of clot formation which can lead to thrombotic events. Antiplatelet agents have been found to reduce cardiovascular events in different clinical settings. The commonest agent that has been used is aspirin which works by inhibiting the cyclooxygenase pathway within the platelet and consequently preventing the release of tromboxane A2. A second group of agents called thienopyridines can inhibit platelets by blocking the P2Y12 receptor. Clopidogrel (Plavix) is currently a widely used thienopyridine that has been used for the treatment of patients presenting with the acute coronary syndrome and patients undergoing percutaneous coronary angioplasty (PCI). Antiplatelet therapy has reduced the occurrence of thrombotic events following PCI, including myocardial infarction and stent thrombosis. However, despite dual therapy with aspirin and clopidogrel, a significant number of patients continue to experience cardiovascular events. There is a now growing body of evidence that recurrence of ischemic complications may be attributed to poor response to clopidogrel and that persistence of enhanced platelet reactivity despite the use of clopidogrel is believed to be clinically relevant.1 The mechanisms leading to poor clopidogrel effects are not fully explained.

Our pilot study will use the VerifyNow device as an ex vivo method to measure platelet inhibition in patients treated with clopidogrel in the setting of STEMI. Since July 2004, the standard of care at the University of Ottawa Heart Institute for the treatment of STEMI has been primary PCI in which all patients receive aspirin 160 mg po either in the field or on arrival in the emergency department and clopidogrel 600 mg po given on arrival to the hospital. Little is known of the pharmacokinetics of clopidogrel in the setting of STEMI. Clopidogrel must be absorbed and activated by the liver to be effective. The physiological mechanisms for these steps may be greatly disturbed in patients presenting with STEMI. Therefore, the purpose of this study will be to examine the degree of platelet inhibition at various time points in this select patient population using the current 600 mg dose of clopidogrel and comparing this dose to other doses of clopidogrel to determine the optimal loading dose in the context of STEMI.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic chest discomfort of greater than 30 minutes duration
2. Onset of chest pain less than 12 hrs prior to entry into the study
3. ST segment elevation of > 1 mm (0.1 mV) in two or more contiguous electrocardiographic leads (on a standard 12 lead ECG) or left bundle branch block not known to be old

Exclusion Criteria:

1. Active bleeding
2. GI or GU bleed within 2 weeks, or any major bleeding episode within 2 weeks
3. Stroke within 90 days or intracranial bleeding at any time
4. Major surgery or trauma within the past six weeks
5. Uncontrolled hypertension (SBP > 200 mm Hg and/or DBP > 110 mm Hg despite treatment)
6. Prolonged (>10 min) cardiopulmonary resuscitation
7. Inadequate vascular access
8. PCI within the last 30 days
9. Thrombolytic agents within the preceding 7 days
10. GP IIb/IIIa antagonists within the preceding 7 days
11. Coagulation disorder (i.e. INR >2.0, platelets <100,000 / mm3, or hematocrit <30%)
12. Current warfarin treatment
13. A subcutaneous therapeutic dose of any LMWH within 12 hours
14. Intolerance to aspirin or clopidogrel
15. Patient already on chronic clopidogrel therapy
16. Other medical condition that is likely to result in death within 12 months
17. Participation in a study with another investigational device or drug < four weeks
18. Pregnancy
19. Known severe renal impairment (creatinine clearance rate of less than 30 ml per minute)
20. Sustained hypotension defined as SBP < 80 mmHg or the need for IV inotropes and/or intraaortic balloon counterpulsation to support the blood pressure
21. Known severe contrast (dye) allergy
22. Inability to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of this randomized pilot study is to evaluate the inhibition of platelet aggregation (IPA) amongst 4 different loading doses of clopidogrel in patients with STEMI treated with bivalirudin as anticoagulant for PCI | Up to 48hrs

SECONDARY OUTCOMES:
Clinical events (death reinfarction, stroke, bleeding) | Up to 6 months
The percent TIMI grade 3 coronary flow at first contrast injection on the base-line angiogram, to TIMI flow after the PCI, | Pre and post ballon injection

CONTACTS AND LOCATIONS:
Overall Officials: Michel R Le May, MD FRCPC FACC, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada